CLINICAL TRIAL: NCT05790811
Title: Validation of Hand & Wrist Physical Exam Video Aid for Improvement of Patient Comprehension
Brief Title: Engaging Patients for Physical Exams During Virtual Care Visits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Charles S Day, Interim Chairman & Medical Director, Professor of Orthopaedic Surgery, Department of Orthopaedic Surgery & Service Line, Wayne State University School of Medicine, Henry Ford Health, Henry Ford Health System
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 14760
Record Dates: First submitted 2023-01-19; First posted 2023-03-30 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Self-preformed Hand Examination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient-oriented video (Experimental): A patient-oriented video with the goal of instructing patients about the maneuvers needed to make specific diagnoses of the hand and wrist. Wording was changed so that it was more patient friendly and text was added to the screen.
  Interventions: Other: Patient-oriented video
- physician-oriented training video (Active Comparator): A physician-oriented video with the goal of instructing physicians on the maneuvers needed to make specific diagnoses of the hand and wrist.
  Interventions: Other: Physician-oriented Video

INTERVENTIONS:
Other: Physician-oriented Video — previously validated Hand and Wrist Examination Video by NEJM designed for usage by a physician in diagnosing common hand and wrist diagnoses
  Arms: physician-oriented training video
Other: Patient-oriented video — The previously validated Hand and Wrist Examination Video by NEJM was modified via the "TogoTiki" application and approved by a patient advisory council.
  Arms: patient-oriented video

SUMMARY:
The goal of this clinical trial is to validate patient-oriented edits to a guided video on self-performed hand examination in participants with no prior hand diagnoses or medical background. The study aims to:

* examine the effect of adding interactive components to an existing orthopedic provider video
* determine if these changes enhance patients' understanding of hand and wrist anatomy as well as carpal tunnel syndrome
* determine if patients are able to use this video to perform an effective physical exam Participants will watch an original physician-oriented training video and a second version (patient-oriented video), which was edited with the input of a patient advisory committee to include interactive elements and a slower speed. The order in which the participants will watch the video will be randomized.

If there is a comparison group: Researchers will compare knowledge scores and general patient preference between the two videos being examined.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age
* Patients who comprehend and speak English
* Patients with carpal tunnel syndrome confirmed on EMG and/or symptoms consistent with carpal tunnel syndrome, including bilateral hand pain, non-traumatic hand pain, and/or numbness/tingling in hand.

Exclusion Criteria:

* Patients under 18 years of age
* Patients who do not speak or comprehend English
* Patients who have cognitive impairments that would be detrimental to understanding of video
* Patients whose symptoms do not match carpal tunnel syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Knowledge Score immediately following the viewing of a video presenting the knowledge | 10 minutes after viewing the video
  Score of the quiz examining the understanding of the contents of the video by the participants. Scoring was a likert scale of 1-5 where 5 represented easy to understand and 1 was very difficult to understand. Separate questions scored as a 1 or 0 where 1 equated to answering the knowledge question correctly and 0 was answering the question incorrectly.

SECONDARY OUTCOMES:
Knowledge Score immediately prior to the viewing of a video presenting the knowledge | 10 minutes before viewing the video
  Score of the quiz examining the participants' understanding prior to watching the video. Scoring was a likert scale of 1-5 where 5 represented easy to understand and 1 was very difficult to understand. Separate questions scored as a 1 or 0 where 1 equated to answering the knowledge question correctly and 0 was answering the question incorrectly.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided